CLINICAL TRIAL: NCT00388765
Title: Protocol to Establish a Research Sample Bank of Lung Biopsy and BAL Samples for a Non-Atopic, Non-Asthmatic Subject Cohort
Brief Title: Normal Control Cohort Sample Bank
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: H-2006-0240
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bronchoscopy; sample bank; research study volunteer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is designed to collect lung washing samples and small pieces of tissue (biopsies) from the lungs of people who do not have any allergies or asthma. These samples will be used by researchers in the future as control samples to compare to samples from people with chronic lung diseases such as allergic asthma or emphysema. Control samples are samples are very important in laboratory experiments so that the researchers can tell what may be labeled as different or abnormal in samples from people with lung disease.

DETAILED DESCRIPTION:
Participants in this study must be between the ages of 18 and 45 years and have no general health concerns and do not have allergies or asthma. If qualified, participants will come to the study site up to 3 times over about a 3-week period. This study involves answering questions about your medical history, having a physical exam, urine pregnancy tests for females who might be able to have children, and breathing tests. You will also have a blood draw to test for bleeding problems and an allergy skin test to see if you are allergic to common things. If it is safe for you, you will have a bronchoscopy. A bronchoscopy is a medical procedure to get samples of cells and small pieces of tissue (biopsies) from your lungs.

The study has some risks. The breathing tests may cause you to feel short of breath or dizzy. The allergy skin test will itch and cause a reaction like a mosquito bite.

There are some risks involved with the bronchoscopy. Most people get a sore throat and feel tired after the procedure. You may need to feel a little short of breath. There is a very rare risk of serious problems.

Women are able to join this study only if they are not pregnant or breast-feeding. If you have plans to become pregnant during the time period in which the study takes place, you should not join this study. For women, a urine pregnancy test will be done at the first visit and you will be asked to be on birth control. The study staff can talk to you about the type of birth control that is all right to use in this study.

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible for participation in the study if all of the following criteria apply:

  * Ability to give a valid informed consent to participate by signing and dating a written consent form.
  * Male or female with no chronic or acute health concerns that might affect subject safety during the study or interfere with the study results, 18-45 years of age
  * An FEV1 > 80% of predicted with an FEV1/FVC ratio above 0.70
  * Methacholine PC20 >16 mg/ml
  * Skin test negative to panel of 12 common aeroallergens

Exclusion Criteria:

* A subject is not eligible to participate in this study if any of the following criteria apply:

  * Medications other than for contraception or OTC pain medications to be approved by PI
  * Recent smoker (within 5 years) or has a smoking history exceeding 5 pack years
  * Currently participating in another clinical trial or has participated in an investigational drug trial with in one month of the screening visit
  * Unable, in the judgment of the investigator, to comply with directions and/or tolerate the procedures required for participation in this trial,
  * Pregnant or breast-feeding or has a planned pregnancy during the course of the study
  * History of bleeding with trauma or abnormal clotting tests
  * History of allergy to any of the medications/sedatives that may be administered during the bronchoscopy procedure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar N Jarjour, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States